CLINICAL TRIAL: NCT04003155
Title: A Phase 3, Randomized, Placebo-controlled, 12-week Double-blind Study, Followed by a Non-Controlled Extension Treatment Period, to Assess the Efficacy and Safety of Fezolinetant in Women Suffering From Moderate to Severe Vasomotor Symptoms (Hot Flashes) Associated With Menopause
Brief Title: A Study to Find Out if Fezolinetant Helps Reduce Moderate to Severe Hot Flashes in Women Going Through Menopause
Acronym: Skylight 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2693-CL-0301; 2018-003528-35 (EudraCT Number)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2022-08-12 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Hot Flashes
Keywords: menopause; ESN364; vasomotor symptoms; fezolinetant
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Double-blind Period: Placebo (Placebo Comparator): Participants received fezolinetant matching placebo (two fezolinetant matching placebo tablets) orally, once daily (QD) up to week 12 during double-blind treatment period.
  Interventions: Drug: placebo
- Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg (Experimental): Participants received fezolinetant 30 mg (one 30 mg fezolinetant tablet and one placebo tablet) orally, QD up to week 12 during double-blind treatment period followed by fezolinetant 30 mg orally, QD from week 13 up to Week 52 during extension treatment period.
  Interventions: Drug: fezolinetant
- Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg (Experimental): Participants received fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD up to week 12 during double-blind treatment period followed by fezolinetant 45 mg orally, QD from week 13 up to Week 52 during extension treatment period.
  Interventions: Drug: fezolinetant
- Double-blind Period: Placebo /Extension Period: Fezolinetant 30 mg (Experimental): Participants who received placebo during double-blind treatment period were re-randomized to receive fezolinetant 30 mg orally, QD from week 13 up to week 52 during extension treatment period.
  Interventions: Drug: fezolinetant
- Double-blind Period: Placebo /Extension Period: Fezolinetant 45 mg (Experimental): Participants who received placebo during double-blind treatment period were re-randomized to receive fezolinetant 45 mg orally, QD from week 13 up to week 52 during extension treatment period.
  Interventions: Drug: fezolinetant

INTERVENTIONS:
Drug: fezolinetant — Oral Tablet
  Arms: Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg; Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg; Double-blind Period: Placebo /Extension Period: Fezolinetant 30 mg; Double-blind Period: Placebo /Extension Period: Fezolinetant 45 mg
Drug: placebo — Oral Tablet
  Arms: Double-blind Period: Placebo

SUMMARY:
This study was for women in menopause with moderate to severe hot flashes. Menopause, a normal part of aging, is the time of a woman's last period. Hot flashes can interrupt a woman's daily life. The study treatments were fezolinetant 30 milligrams (mg) (1 tablet of fezolinetant and 1 placebo tablet) once a day, fezolinetant 45 mg (2 tablets of fezolinetant) once a day or placebo (2 tablets) once a day. (Placebo was a dummy treatment that looks like medicine but did not had any medicine in it.) The study compared fezolinetant and placebo after 4 and 12 weeks of dosing. The study evaluated if fezolinetant reduces the number of hot flashes. And the study evaluated if fezolinetant reduces the severity of the hot flashes. Women in the study received an electronic handheld device at the first study visit. (It was similar to a smart phone.) Each day of the study, study participants used this to record their hot flashes. Their record for the 10 days before the start of study treatment was checked. They remained in the study if their record shown 7 or 8 moderate to severe hot flashes per day (50 or more per week). Next, they were picked for 1 of the 2 study treatments (fezolinetant or placebo) by chance alone. It was like flipping a coin. The study participants took study treatment for 52 weeks. The first 12 weeks of study treatment are "double-blinded." That means that the study participants and the study doctors did not knew who took which of the study treatments (fezolinetant 30 mg, fezolinetant 45 mg or placebo) during that time. The last 40 weeks of study treatment are "noncontrolled." That means that each study participant and the study doctors knew which study treatment that study participant took during that time. Women who took fezolinetant during the first 12 weeks continued to take the same dose. Women who took placebo during the first 12 weeks took fezolinetant. Their dose was either 30 mg or 45 mg fezolinetant. At weeks 2, 4, 8, 12, 14, 16 and then once a month, the study participants visited the hospital or clinic for a check-up. They were asked about medications, side effects and how they felt. Other checks included physical exam and vital signs (heart rate, temperature and blood pressure). Blood and urine was collected for laboratory tests. Study participants completed questionnaires that were about how hot flashes affect their daily life. Study participants who still had their uterus had the following 2 tests done at the first and last study visits. One of the 2 tests was endometrial biopsy. This test involves removing a small amount of tissue from the inside lining of the uterus. The tissue was then checked under a microscope. The other test is transvaginal ultrasound. This test used sound waves to create pictures of the organs in the pelvis. The sound waves were transmitted by a probe (transducer), which was placed inside the vagina. Study participants may have a screening mammogram done at the first and/or last study visit. A mammogram is an x-ray picture of the breasts used to screen for breast cancer. Study participants who did not had this test done in the last 12 months had it done at the first study visit. They had it done at the last study visit if they are due for their screening mammogram and their own doctor agrees. The last check-up at the hospital or clinic was 3 weeks after the last dose of study treatment.

DETAILED DESCRIPTION:
This study consisted of a screening period and a 52 week treatment period. Safety follow up occurred 3 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index ≥ 18 kg/m^2 and ≤ 38 kg/m^2.
* Subject must be seeking treatment or relief for vasomotor symptoms (VMS) associated with menopause and confirmed as menopausal per 1 of the following criteria at the screening visit:

  * Spontaneous amenorrhea for ≥ 12 consecutive months
  * Spontaneous amenorrhea for ≥ 6 months with biochemical criteria of menopause (follicle-stimulating hormone [FSH] > 40 IU/L); or
  * Having had bilateral oophorectomy ≥ 6 weeks prior to the screening visit.
* Within the 10 days prior to randomization, subject must have a minimum average of 7 to 8 moderate to severe hot flashes (HFs) vasomotor symptoms (VMS) per day, or 50 to 60 per week.
* Subject is in good general health as determined on the basis of medical history and general physical examination, including a bimanual clinical pelvic examination and clinical breast examination devoid of relevant clinical findings, performed at the screening visit; hematology and biochemistry parameters, pulse rate and/or blood pressure and electrocardiogram (ECG) within the reference range for the population studied, or showing no clinically relevant deviations.
* Subject has documentation of a normal/negative or no clinically significant findings mammogram (obtained at screening or within the prior 12 months of study enrollment). Appropriate documentation includes a written report or an electronic report indicating normal/negative or no clinically significant mammographic findings.
* Subject is willing to undergo a transvaginal ultrasound (TVU) to evaluate the uterus and ovaries at screening and at week 52 end of treatment (EOT), and for subjects who are withdrawn from the study prior to completion, a TVU at the early discontinuation (ED) visit.
* Subject is willing to undergo an endometrial biopsy at screening and at week 52 (EOT), for subjects with uterine bleeding, and for subjects who are withdrawn from the study prior to completion. The endometrial biopsy obtained at screening must be considered evaluable.
* Subject has documentation of a normal or not clinically significant Papanicolaou (Pap) test (or equivalent cervical cytology) within the previous 12 months or at screening.
* Subject has a negative urine pregnancy test at screening.
* Subject has a negative serology panel (i.e., negative hepatitis B surface antigen, negative hepatitis C virus antibody and negative human immunodeficiency virus antibody screens) at screening.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject uses a prohibited therapy (strong or moderate cytochrome P450 1A2 [CYP1A2] inhibitors, hormone replacement therapy [HRT], hormonal contraceptive or any treatment for VMS [prescription, over the counter or herbal]) or is not willing to wash out and discontinue use of such drugs for the full duration of study conduct.
* Subject has known substance abuse or alcohol addiction within 6 months of screening.
* Subject has previous or current history of a malignant tumor, except for basal cell carcinoma.
* Subject's systolic blood pressure is ≥ 130 mmHg or diastolic blood pressure is ≥ 80 mmHg based on the average of 2 to 3 readings, on at least 2 different occasions within the screening period.

  * Subjects who do not meet these criteria may be re-assessed after initiation or review of antihypertensive measures.
  * Subjects with a medical history of hypertension can be enrolled once they are medically clear (stable and compliant).
* Subject has history of severe allergy, hypersensitivity or intolerance to drugs in general, including the study drug and any of its excipients.
* Subject has an unacceptable result from the TVU assessment at screening (i.e., full length of endometrial cavity cannot be visualized or presence of a clinically significant finding).
* Subject has an endometrial biopsy confirming presence of disordered proliferative endometrium, endometrial hyperplasia, endometrial cancer or other clinically significant findings at screening.
* Subject has a history within the last 6 months of undiagnosed uterine bleeding.
* Subject has a history of seizures or other convulsive disorders.
* Subject has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Subject has active liver disease, jaundice or elevated liver aminotransferases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]), elevated total or direct bilirubin, elevated international normalized ratio (INR), or elevated alkaline phosphatase (ALP). Patients with mildly elevated ALT or AST up to 1.5 times the upper limit of normal (ULN) can be enrolled if total and direct bilirubin are normal. Patients with mildly elevated ALP (up to 1.5 x ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Patients with Gilbert's syndrome with elevated total bilirubin may be enrolled as long as direct bilirubin, hemoglobin and reticulocytes are normal.
* Subject has creatinine > 1.5 × ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease formula ≤ 59 mL/min per 1.73 m^2 at screening.
* Subject has a history of suicide attempt or suicidal behavior within the last 12 months or has suicidal ideation within the last 12 months (a response of "yes" to question 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale [C-SSRS]), or who is at significant risk to commit suicide at screening and at randomization.
* Subject has previously been enrolled in a clinical trial with fezolinetant.
* Subject is participating concurrently in another interventional study or participated in an interventional study within 28 days prior to screening, or received any investigational drug within 28 days or within 5 half-lives prior to screening, whichever is longer.
* Subject is unable or unwilling to complete the study procedures.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has had partial or full hysterectomy.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (95):
- United States (71):
  - SEC Clinical Research, Andalusia, Alabama
  - Central Research Associates, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Ensley, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Advanced Clinical Research - Rancho Paseo, Banning, California
  - Hope Clinical Research, LLC, Canoga Park, California
  - Alliance Research Inc, Canoga Park, California
  - Marvel Clinical Research, Huntington Beach, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - National Research Institute - Panorama, Los Angeles, California
  - Northern California Research, Sacramento, California
  - Precision Research Institute, Inc, San Diego, California
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Precision Clinical Research, Coral Springs, Florida
  - American Research Institute, Inc., Cutler Bay, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Vital Pharma Research Inc., Hialeah, Florida
  - Health Awareness, Jupiter, Florida
  - GYN Research Center, Kissimmee, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Altus Research, Lake Worth, Florida
  - Medical Research Center of Miami II, Miami, Florida
  - Spotlight research center, Miami, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Cornerstone Research Institute, Orlando, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - Health Awareness, Port Saint Lucie, Florida
  - International Clinical Research, Sanford, Florida
  - Premier Medical Associates, The Villages, Florida
  - Better Health Greater Life, Atlanta, Georgia
  - Gwinnett Research Institute, Buford, Georgia
  - IACT Health, Columbus, Georgia
  - NuDirections Clinical Research, Duluth, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - The Healing Sanctuary, LLC, Idaho Falls, Idaho
  - Avant Research Associates, LLC, Crowley, Louisiana
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Saginaw Valley Medical Research Group, Llc, Saginaw, Michigan
  - Montana Medical Research Inc, Missoula, Montana
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Office Of Edmond Pack, Md, Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - Unified Women's Clinical Research, Greensboro, North Carolina
  - Unified Womens Clinical Research, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Unified Women's Clinical Research, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Velocity Clinical Research, Cincinnati, Ohio
  - Complete Healthcare For Women, Columbus, Ohio
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Invocare Clinical Research Center, West Columbia, South Carolina
  - Medical Research Center of Memphis LLC, Memphis, Tennessee
  - International Clinical Research, Murfreesboro, Tennessee
  - Accent Clinical Research Professionals, Allen, Texas
  - DiscoveResarch, Inc., Bryan, Texas
  - Protenium Clinical Research, LLC, Hurst, Texas
  - EPIC Medical Research, Murray, Utah
  - Tidewater Clinical Research, Inc., Virginia Beach, Virginia
- Canada (5):
  - Site CA15003, Brampton, Ontario
  - Site CA15002, Point Claire, Quebec
  - Site CA15001, Québec, Quebec
  - Site CA15004, Québec, Quebec
  - Site CA15006, Québec, Quebec
- Czechia (2):
  - Site CZ42003, Vodňany, Jihočeský kraj
  - Site CZ42001, Olomouc
- Hungary (3):
  - Site HU36004, Debrecen
  - Site HU36001, Kecskemét
  - Site HU36002, Szekesfeherver
- Poland (9):
  - Site PL48012, Katowice, Silesian Voivodeship
  - Site PL48003, Bialystok
  - Site PL48013, Katowice
  - Site PL48004, Katowice
  - Site PL48007, Lublin
  - Site PL48005, Poznan
  - Site PL48014, Świdnik
  - Site PL48009, Warsaw
  - Site PL48001, Warsaw
- Site ES34004, Seville, Spain
- United Kingdom (4):
  - Site GB44001, Wokingham, Berkshire
  - Site GB44003, Orpington, Kent
  - Site GB44002, Coventry, Warwickshire
  - Site GB44004, Middlesex

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Shapiro C M M, Neal-Perry G, Stute P, Thurston RC, Wolfman W, English M, Wu X, Ottery FD. Early onset, maintenance of effect, and day-/night-time findings following fezolinetant treatment for moderate to severe vasomotor symptoms associated with menopause: A pooled phase 3 analysis. Maturitas. 2025 Dec;203:108740. doi: 10.1016/j.maturitas.2025.108740. Epub 2025 Oct 6. PMID 41259888
- [Derived] Santoro N, Neal-Perry G, Stute P, Blogg M, Mancuso S, Morga A, Ottery FD, Siddiqui E. Fezolinetant effect on vasomotor symptoms due to menopause in women unsuitable for hormone therapy. Curr Med Res Opin. 2025 Feb;41(2):375-384. doi: 10.1080/03007995.2025.2470752. Epub 2025 Mar 5. PMID 40044127
- [Derived] Kagan R, Cano A, Nappi RE, English ML, Mancuso S, Wu X, Ottery FD. Safety of Fezolinetant for Treatment of Moderate to Severe Vasomotor Symptoms Due to Menopause: Pooled Analysis of Three Randomized Phase 3 Studies. Adv Ther. 2025 Feb;42(2):1147-1164. doi: 10.1007/s12325-024-03073-8. Epub 2024 Dec 30. PMID 39739195
- [Derived] Morga A, Zimmermann L, Valluri U, Siddiqui E, McLeod L, Bender RH. Validation and Application of Thresholds to Define Meaningful Change in Vasomotor Symptoms Frequency: Analysis of Pooled SKYLIGHT 1 and 2 Data. Adv Ther. 2024 Jul;41(7):2845-2858. doi: 10.1007/s12325-024-02849-2. Epub 2024 May 22. PMID 38775925
- [Derived] Schultz NM, Morga A, Siddiqui E, Rhoten SE. Psychometric Evaluation of the MENQOL Instrument in Women Experiencing Vasomotor Symptoms Associated with Menopause. Adv Ther. 2024 Jun;41(6):2233-2252. doi: 10.1007/s12325-024-02787-z. Epub 2024 Feb 24. PMID 38396203
- [Derived] Schultz NM, Morga A, Siddiqui E, Rhoten SE. Psychometric evaluation of the PROMIS SD-SF-8b instrument in individuals experiencing vasomotor symptoms due to menopause. Health Qual Life Outcomes. 2023 Nov 21;21(1):126. doi: 10.1186/s12955-023-02206-x. PMID 37990323
- [Derived] O'Malley PA. A Nonhormonal Selective NK3R Antagonist for Moderate to Severe Vasomotor Symptoms in Menopause. Clin Nurse Spec. 2023 Nov-Dec 01;37(6):259-261. doi: 10.1097/NUR.0000000000000774. No abstract available. PMID 37870510
- [Derived] Lederman S, Ottery FD, Cano A, Santoro N, Shapiro M, Stute P, Thurston RC, English M, Franklin C, Lee M, Neal-Perry G. Fezolinetant for treatment of moderate-to-severe vasomotor symptoms associated with menopause (SKYLIGHT 1): a phase 3 randomised controlled study. Lancet. 2023 Apr 1;401(10382):1091-1102. doi: 10.1016/S0140-6736(23)00085-5. Epub 2023 Mar 13. PMID 36924778
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14542&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women participants 40 to 65 years of age who had moderate to severe vasomotor symptoms (VMS) and seeking treatment or relief for VMS associated with menopause, confirmed as menopausal, had to have minimum average of 7 to 8 moderate to severe hot flashes (HFs) (VMS) per day within the 10 days prior to randomization and who met the inclusion criteria and none of the exclusion criteria were enrolled in this study.
Pre-assignment Details: Prior to randomization, participants had a screening period during which a minimum 10-day collection of baseline VMS frequency and severity assessments were performed.
Groups:
- Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg: Participants received fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD up to week 12 during double-blind treatment period followed by fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD from week 13 up to week 52 during extension treatment period.
- Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg: Participants who received placebo during double-blind treatment period were re-randomized to receive fezolinetant 30 mg orally, QD from week 13 up to week 52 during extension treatment period.
- Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg: Participants who received placebo during double-blind treatment period were re-randomized to receive fezolinetant 45 mg orally, QD from week 13 up to week 52 during extension treatment period.
Period: Double-Blind (DB) Period (12 Weeks)
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Started | 175 | 176 | 176 | 0 | 0
Full Analysis Set | 175 | 173 | 174 | 0 | 0
Safety Analysis Set | 175 | 174 (1 participant who was randomized to fezolinetant 45 mg received fezolinetant 30 mg during the 12-week study period. This participant was included in the fezolinetant 30 mg group for the Safety Analysis Set) | 173 | 0 | 0
Treated | 175 | 173 | 174 (1 participant who was randomized in this arm actually received 30mg fezolinetant.) | 0 | 0
Completed | 152 | 142 | 161 | 0 | 0
Not Completed | 23 | 34 | 15 | 0 | 0
Not completed — Adverse Event | 9 | 8 | 5 | 0 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 3 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 12 | 4 | 0 | 0
Not completed — Miscellaneous | 1 | 7 | 3 | 0 | 0
Period: Extension Period (EP) (40 Weeks)
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Started | 0 (Participants who received placebo in double-blind period were moved to fezolinetant 30/45 mg arms in extension treatment period) | 142 (1 participant who completed DB discontinued study before entering EP. 1 participant who was randomized to 45 mg but received 30 mg in DB, was then moved to 30mg in EP.) | 158 (Two participants who completed double-blind period discontinued the study before entering the extension treatment period) | 76 (Participants who received placebo in double-blind period were randomized to fezolinetant 30 mg arms) | 76 (Participants who received placebo in double-blind period were randomized to fezolinetant 45 mg arms)
Completed | 0 | 124 | 143 | 62 | 67
Not Completed | 0 | 18 | 15 | 14 | 9
Not completed — Adverse Event | 0 | 5 | 4 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 12 | 7 | 9 | 5
Not completed — Miscellaneous | 0 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Double-blind Period: Placebo: Participants received fezolinetant matching placebo (two fezolinetant matching placebo tablets) orally, QD up to week 12 during double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Total
Number analyzed (Participants) | 175 | 176 | 176 | 527
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (4.8) | 54.1 (4.9) | 54.3 (5.2) | 54.4 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 176 | 176 | 527
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 43 | 48 | 137
  Not Hispanic or Latino | 128 | 133 | 128 | 389
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Race: White | 142 | 150 | 143 | 435
  Race: Black or African American | 28 | 21 | 27 | 76
  Race: American Indian or Alaska Native | 2 | 0 | 1 | 3
  Race: Asian | 3 | 3 | 3 | 9
  Race: Pacific Islander | 0 | 0 | 1 | 1
  Race: More Than One Race | 0 | 1 | 1 | 2
  Race: Unknown | 0 | 1 | 0 | 1
Frequency of Moderate and Severe Vasomotor Symptoms per 24 hours [Mean (Standard Deviation); unit: VMS per day] — The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. Baseline was the average number of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization. Population: Full analysis set (FAS) consisted of all participants who were randomized and received at least 1 dose of study intervention. The randomized treatment for each participant was used for summaries by treatment group based on the FAS, even if a participant erroneously received a different treatment.
  VMS per day
    number analyzed (Participants) | 175 | 173 | 174 | 522
    (all) | 10.51 (3.79) | 10.65 (4.73) | 10.44 (3.92) | 10.53 (4.16)
Severity of Moderate and Severe Vasomotor Symptoms per 24 hours [Mean (Standard Deviation); unit: Score on a scale] — Severity of moderate to severe VMS per day was calculated as follows: [(number of moderate VMS × 2) + (number of severe VMS × 3)]/number of daily moderate/severe VMS. Higher score indicates greater severity. Baseline was the weighted average of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization. Population: FAS Population
  Score on a scale
    number analyzed (Participants) | 175 | 173 | 174 | 522
    (all) | 2.43 (0.35) | 2.39 (0.34) | 2.40 (0.35) | 2.41 (0.35)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in The Mean Frequency of Moderate to Severe VMS at Week 4
Description: The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. A daily frequency per week was derived by taking the mean of the data over 7 days. Moderate VMS was defined as sensation of heat with sweating/dampness, but participant was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). Baseline was the average number of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization.
Time Frame: Baseline and week 4
Population: Full analysis set (FAS) consisted of all participants who were randomized and received at least 1 dose of study intervention. The randomized treatment for each participant was used for summaries by treatment group based on the FAS, even if a participant erroneously received a different treatment. Participants with available data at specified time point were included.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Groups:
- Double-blind Period: Fezolinetant 30 mg: Participants received fezolinetant 30 mg (one 30 mg fezolinetant tablet and one placebo tablet) orally, QD up to week 12 during double-blind treatment.
- Double-blind Period: Fezolinetant 45 mg: Participants received fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD up to week 12 during double-blind treatment period.
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 166 | 157 | 164
VMS per day | -3.32 (0.29) | -5.19 (0.30) | -5.39 (0.30)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Least squares Mean (LSM), Standard error (SE), Confidence interval (CI), Mixed model repeated measures (MMRM), Change from Baseline (CFB), Dependent variable (dv), Treatment (tr), Week (wk), Baseline (bl), Weight (wt); Test type: Superiority; p < 0.001, MMRM — LSM, SE, CI, & p-values come from MMRM analysis of covariance model with CFB as dv & trt group, wk & smoking status as factors, with bl measurement & bl wt as covariates, as well as an interaction of trt by wk & interaction of bl measurement by wk; LSMean Difference = -1.87, 95% CI [-2.69 to -1.05], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.07, 95% CI [-2.89 to -1.25], Standard Error of Mean 0.42
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.012, Hochberg
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.007, Hochberg

2. Primary Outcome: Change From Baseline in The Mean Frequency of Moderate to Severe VMS at Week 12
Description: as for outcome 1
Time Frame: Baseline and week 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 139 | 131 | 146
VMS per day | -3.90 (0.31) | -6.28 (0.32) | -6.44 (0.31)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.39, 95% CI [-3.25 to -1.52], Standard Error of Mean 0.44
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.55, 95% CI [-3.40 to -1.70], Standard Error of Mean 0.43
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.012, Hochberg
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.007, Hochberg

3. Primary Outcome: Change From Baseline in The Mean Severity of Moderate to Severe VMS at Week 4
Description: Severity of moderate to severe VMS per day at post baseline visit was calculated as follows:
  [(number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3)]/Total number of daily mild/moderate/severe hot flashes Moderate VMS was defined as sensation of heat with sweating/dampness, but participant was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed).
  Severity was zero for participants that had no mild or moderate or severe VMS. Higher scores indicates greater severity.
Time Frame: Baseline and week 4
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 166 | 157 | 164
Score on a scale | -0.27 (0.04) | -0.42 (0.04) | -0.46 (0.04)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.012, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.15, 95% CI [-0.27 to -0.03], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.19, 95% CI [-0.30 to -0.07], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.012, Hochberg
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.007, Hochberg

4. Primary Outcome: Change From Baseline in The Mean Severity of Moderate to Severe VMS at Week 12
Description: as for outcome 3
Time Frame: Baseline and week 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 139 | 131 | 146
Score on a scale | -0.37 (0.05) | -0.60 (0.05) | -0.57 (0.05)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.24, 95% CI [-0.39 to -0.09], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.007, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.20, 95% CI [-0.35 to -0.06], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.012, Hochberg
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.007, Hochberg

5. Secondary Outcome: Change From Baseline in The Mean Patient-reported Outcomes Measurement Information System Sleep Disturbance - Short Form 8b (PROMIS SD SF 8b) Total Score at Week 12
Description: The PROMIS SD SF 8b assesses self-reported sleep disturbance over the past 7 days and includes perceptions of restless sleep; satisfaction with sleep; refreshing sleep; difficulties sleeping, getting to sleep or staying asleep; amount of sleep; and sleep quality. Because it assesses the participants experience of sleep disturbance, the measure does not focus on specific sleep-disorder symptoms or ask patients to report objective measures of sleep (e.g., total amount of sleep, time to fall asleep and amount of wakefulness during sleep). Responses to each of the 8 items range from 1 (no disturbed sleep) to 5 (disturbed sleep), and the range of possible summed raw scores is 8 to 40. Higher scores on the PROMIS SD SF 8b indicate more of the disturbed sleep.
Time Frame: Baseline and week 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 148 | 133 | 156
Score on a scale | -3.2 (0.5) | -3.7 (0.6) | -4.2 (0.5)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.489, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.5, 95% CI [-2.0 to 1.0], Standard Error of Mean 0.8
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.155, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -1.1, 95% CI [-2.5 to 0.4], Standard Error of Mean 0.7

6. Secondary Outcome: Change From Baseline in The Mean Frequency of Moderate, and Severe VMS to Each Study Week Up to Week 12
Description: as for outcome 1
Time Frame: Baseline and weeks 1, 2, 3, 5, 6, 7, 8, 9, 10 and 11
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 174 | 169 | 166
VMS per day
  Week 1 | -1.82 (0.26) | -3.63 (0.26) | -3.07 (0.26)
  Week 2: number analyzed (Participants) | 171 | 162 | 166
  Week 2 | -2.76 (0.28) | -4.73 (0.28) | -4.58 (0.28)
  Week 3: number analyzed (Participants) | 165 | 159 | 166
  Week 3 | -3.15 (0.28) | -5.14 (0.29) | -5.25 (0.29)
  Week 5: number analyzed (Participants) | 158 | 151 | 159
  Week 5 | -3.49 (0.28) | -5.56 (0.29) | -5.67 (0.29)
  Week 6: number analyzed (Participants) | 156 | 144 | 157
  Week 6 | -3.58 (0.29) | -5.70 (0.30) | -5.97 (0.29)
  Week 7: number analyzed (Participants) | 154 | 144 | 162
  Week 7 | -3.71 (0.30) | -5.80 (0.31) | -5.97 (0.30)
  Week 8: number analyzed (Participants) | 152 | 143 | 151
  Week 8 | -3.71 (0.30) | -6.10 (0.31) | -6.10 (0.30)
  Week 9: number analyzed (Participants) | 148 | 141 | 152
  Week 9 | -4.09 (0.30) | -6.16 (0.31) | -6.24 (0.30)
  Week 10: number analyzed (Participants) | 141 | 140 | 152
  Week 10 | -4.09 (0.30) | -6.30 (0.31) | -6.25 (0.30)
  Week 11: number analyzed (Participants) | 144 | 138 | 149
  Week 11 | -3.89 (0.31) | -6.37 (0.31) | -6.34 (0.30)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.81, 95% CI 2-sided [-2.53 to -1.09], Standard Error of Mean 0.37
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -1.25, 95% CI 2-sided [-1.97 to -0.53], Standard Error of Mean 0.37
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -1.97, 95% CI 2-sided [-2.75 to -1.19], Standard Error of Mean 0.40
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -1.83, 95% CI 2-sided [-2.60 to -1.05], Standard Error of Mean 0.39
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -1.99, 95% CI 2-sided [-2.79 to -1.19], Standard Error of Mean 0.41
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.10, 95% CI 2-sided [-2.90 to -1.31], Standard Error of Mean 0.40
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.07, 95% CI 2-sided [-2.87 to -1.27], Standard Error of Mean 0.41
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.18, 95% CI 2-sided [-2.98 to -1.39], Standard Error of Mean 0.40
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.11, 95% CI 2-sided [-2.92 to -1.30], Standard Error of Mean 0.41
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.39, 95% CI 2-sided [-3.19 to -1.59], Standard Error of Mean 0.41
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.10, 95% CI 2-sided [-2.95 to -1.25], Standard Error of Mean 0.43
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.27, 95% CI 2-sided [-3.11 to -1.42], Standard Error of Mean 0.43
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.39, 95% CI 2-sided [-3.25 to -1.54], Standard Error of Mean 0.43
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.39, 95% CI 2-sided [-3.23 to -1.55], Standard Error of Mean 0.43
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.08, 95% CI 2-sided [-2.93 to -1.22], Standard Error of Mean 0.43
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.16, 95% CI 2-sided [-3.00 to -1.31], Standard Error of Mean 0.43
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.21, 95% CI 2-sided [-3.05 to -1.37], Standard Error of Mean 0.43
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.16, 95% CI 2-sided [-2.98 to -1.33], Standard Error of Mean 0.42
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.48, 95% CI 2-sided [-3.34 to -1.62], Standard Error of Mean 0.44
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -2.45, 95% CI 2-sided [-3.30 to -1.60], Standard Error of Mean 0.43

7. Secondary Outcome: Change From Baseline in The Mean Severity of Moderate, and Severe VMS to Each Study Week Up to Week 12
Description: as for outcome 3
Time Frame: Baseline and weeks 1, 2, 3, 5, 6, 7, 8, 9, 10 and 11
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 175 | 173 | 174
Score on a scale
  Week 1: number analyzed (Participants) | 174 | 169 | 166
  Week 1 | -0.15 (0.03) | -0.25 (0.03) | -0.25 (0.03)
  Week 2: number analyzed (Participants) | 171 | 162 | 168
  Week 2 | -0.21 (0.03) | -0.35 (0.04) | -0.36 (0.03)
  Week 3: number analyzed (Participants) | 165 | 159 | 166
  Week 3 | -0.27 (0.04) | -0.43 (0.04) | -0.43 (0.04)
  Week 5: number analyzed (Participants) | 158 | 151 | 159
  Week 5 | -0.29 (0.04) | -0.46 (0.04) | -0.46 (0.04)
  Week 6: number analyzed (Participants) | 156 | 144 | 157
  Week 6 | -0.30 (0.05) | -0.50 (0.05) | -0.55 (0.05)
  Week 7: number analyzed (Participants) | 154 | 144 | 162
  Week 7 | -0.28 (0.05) | -0.52 (0.05) | -0.54 (0.05)
  Week 8: number analyzed (Participants) | 152 | 143 | 151
  Week 8 | -0.29 (0.05) | -0.57 (0.05) | -0.53 (0.05)
  Week 9: number analyzed (Participants) | 148 | 141 | 152
  Week 9 | -0.35 (0.05) | -0.62 (0.05) | -0.56 (0.05)
  Week 10: number analyzed (Participants) | 141 | 140 | 152
  Week 10 | -0.34 (0.05) | -0.62 (0.05) | -0.57 (0.05)
  Week 11: number analyzed (Participants) | 144 | 138 | 149
  Week 11 | -0.37 (0.06) | -0.64 (0.06) | -0.61 (0.06)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.10, 95% CI 2-sided [-0.17 to -0.03], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.10, 95% CI 2-sided [-0.17 to -0.03], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.15, 95% CI 2-sided [-0.24 to -0.05], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.15, 95% CI 2-sided [-0.25 to -0.06], Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p = 0.004, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.16, 95% CI 2-sided [-0.27 to -0.05], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.17, 95% CI 2-sided [-0.28 to -0.06], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.17, 95% CI 2-sided [-0.29 to -0.05], Standard Error of Mean 0.06
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p = 0.004, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.17, 95% CI 2-sided [-0.29 to -0.06], Standard Error of Mean 0.06
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.20, 95% CI 2-sided [-0.33 to -0.07], Standard Error of Mean 0.07
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.25, 95% CI 2-sided [-0.38 to -0.13], Standard Error of Mean 0.06
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.24, 95% CI 2-sided [-0.37 to -0.11], Standard Error of Mean 0.07
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.26, 95% CI 2-sided [-0.39 to -0.13], Standard Error of Mean 0.07
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.28, 95% CI 2-sided [-0.41 to -0.15], Standard Error of Mean 0.07
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.24, 95% CI 2-sided [-0.37 to -0.11], Standard Error of Mean 0.07
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; MMRM = -0.26, 95% CI 2-sided [-0.41 to -0.12], Standard Error of Mean 0.07
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p = 0.004, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.21, 95% CI 2-sided [-0.35 to -0.06], Standard Error of Mean 0.07
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.28, 95% CI 2-sided [-0.43 to -0.13], Standard Error of Mean 0.08
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.23, 95% CI 2-sided [-0.37 to -0.08], Standard Error of Mean 0.07
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.27, 95% CI 2-sided [-0.43 to -0.12], Standard Error of Mean 0.08
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -0.24, 95% CI 2-sided [-0.40 to -0.09], Standard Error of Mean 0.08

8. Secondary Outcome: Mean Percent Change in The Frequency of Moderate And Severe VMS From Baseline to Each Study Week Up to Week 12
Description: as for outcome 1
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 175 | 173 | 174
Percent change
  Week 1: number analyzed (Participants) | 174 | 169 | 166
  Week 1 | -16.63 (2.31) | -32.15 (2.34) | -28.84 (2.35)
  Week 2: number analyzed (Participants) | 171 | 162 | 168
  Week 2 | -25.08 (2.50) | -42.37 (2.55) | -43.37 (2.54)
  Week 3: number analyzed (Participants) | 165 | 159 | 166
  Week 3 | -28.81 (2.54) | -46.94 (2.59) | -50.00 (2.57)
  Week 4: number analyzed (Participants) | 166 | 157 | 164
  Week 4 | -30.59 (2.67) | -47.34 (2.72) | -51.65 (2.69)
  Week 5: number analyzed (Participants) | 158 | 151 | 159
  Week 5 | -32.55 (2.65) | -50.12 (2.71) | -54.33 (2.67)
  Week 6: number analyzed (Participants) | 156 | 144 | 157
  Week 6 | -33.35 (2.72) | -51.74 (2.78) | -57.18 (2.73)
  Week 7: number analyzed (Participants) | 154 | 144 | 162
  Week 7 | -34.85 (2.86) | -53.14 (2.93) | -56.26 (2.85)
  Week 8: number analyzed (Participants) | 152 | 143 | 151
  Week 8 | -35.71 (2.83) | -55.88 (2.90) | -56.89 (2.83)
  Week 9: number analyzed (Participants) | 148 | 141 | 152
  Week 9 | -39.64 (2.87) | -56.31 (2.93) | -58.54 (2.85)
  Week 10: number analyzed (Participants) | 141 | 140 | 152
  Week 10 | -39.51 (2.81) | -57.39 (2.87) | -59.01 (2.79)
  Week 11: number analyzed (Participants) | 144 | 138 | 149
  Week 11 | -38.05 (2.84) | -58.37 (2.90) | -60.18 (2.82)
  Week 12: number analyzed (Participants) | 139 | 131 | 146
  Week 12 | -37.06 (2.89) | -57.13 (2.95) | -61.24 (2.86)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -15.52, 95% CI 2-sided [-21.99 to -9.06], Standard Error of Mean 3.29
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -12.22, 95% CI 2-sided [-18.69 to -5.74], Standard Error of Mean 3.30
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -17.30, 95% CI 2-sided [-24.32 to -10.27], Standard Error of Mean 3.57
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -18.29, 95% CI 2-sided [-25.30 to -11.29], Standard Error of Mean 3.57
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -18.13, 95% CI 2-sided [-25.25 to -11.00], Standard Error of Mean 3.63
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -21.19, 95% CI 2-sided [-28.29 to -14.09], Standard Error of Mean 3.61
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 4; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -16.75, 95% CI 2-sided [-24.24 to -9.26], Standard Error of Mean 3.81
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 4; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -21.05, 95% CI 2-sided [-28.50 to -13.61], Standard Error of Mean 3.79
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -17.57, 95% CI 2-sided [-25.02 to -10.12], Standard Error of Mean 3.79
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -21.78, 95% CI 2-sided [-29.18 to -14.39], Standard Error of Mean 3.76
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -18.39, 95% CI 2-sided [-26.03 to -10.75], Standard Error of Mean 3.89
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -23.83, 95% CI 2-sided [-31.39 to -16.27], Standard Error of Mean 3.85
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -18.29, 95% CI 2-sided [-26.33 to -10.25], Standard Error of Mean 4.09
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -21.41, 95% CI 2-sided [-29.35 to -13.48], Standard Error of Mean 4.04
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -20.16, 95% CI 2-sided [-28.14 to -12.19], Standard Error of Mean 4.06
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -21.17, 95% CI 2-sided [-29.04 to -13.30], Standard Error of Mean 4.01
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -16.67, 95% CI 2-sided [-24.73 to -8.61], Standard Error of Mean 4.10
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -18.89, 95% CI 2-sided [-26.84 to -10.94], Standard Error of Mean 4.05
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -17.88, 95% CI 2-sided [-25.77 to -9.99], Standard Error of Mean 4.01
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -19.50, 95% CI 2-sided [-27.28 to -11.72], Standard Error of Mean 3.96
Statistical Analysis 21: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -20.32, 95% CI 2-sided [-28.30 to -12.35], Standard Error of Mean 4.06
Statistical Analysis 22: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -22.14, 95% CI 2-sided [-30.00 to -14.28], Standard Error of Mean 4.00
Statistical Analysis 23: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 12; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -20.08, 95% CI 2-sided [-28.19 to -11.96], Standard Error of Mean 4.13
Statistical Analysis 24: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 12; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -24.18, 95% CI 2-sided [-32.16 to -16.20], Standard Error of Mean 4.06

9. Secondary Outcome: Number of Participants With Percent Reduction of >=50% in the Mean Frequency of Moderate and Severe VMS From Baseline to Each Study Week Up to Week 12
Description: The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. A daily frequency per week was derived by taking the mean of the data over 7 days. Moderate VMS was defined as sensation of heat with sweating/dampness, but participant was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). Baseline was the average number of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization. Participant has >=50% reduction from baseline to each post baseline week for the frequency of moderate to severe VMS.
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: FAS Population
Measure: Number; unit: Participants
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 175 | 173 | 174
Participants
  Week 1 | 18 | 47 | 44
  Week 2 | 37 | 64 | 75
  Week 3 | 42 | 69 | 89
  Week 4 | 49 | 77 | 94
  Week 5 | 47 | 76 | 94
  Week 6 | 50 | 78 | 96
  Week 7 | 52 | 79 | 98
  Week 8 | 52 | 93 | 87
  Week 9 | 56 | 85 | 97
  Week 10 | 45 | 84 | 100
  Week 11 | 55 | 85 | 100
  Week 12 | 52 | 77 | 99
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p < 0.001, Regression, Logistic — Based on logistic regression with treatment group and smoking status (current vs former/never) as factors and mean frequency of vasomotor symptoms at baseline as a covariate; Odds Ratio (OR) = 3.245, 95% CI 2-sided [1.823 to 5.999]
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.964, 95% CI 2-sided [1.658 to 5.497]
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.187, 95% CI 2-sided [1.363 to 3.549]
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.847, 95% CI 2-sided [1.786 to 4.601]
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.096, 95% CI 2-sided [1.326 to 3.345]
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.333, 95% CI 2-sided [2.121 to 5.302]
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 4; Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.061, 95% CI 2-sided [1.323 to 3.233]
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.025, 95% CI 2-sided [1.947 to 4.746]
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.130, 95% CI 2-sided [1.363 to 3.357]
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.223, 95% CI 2-sided [2.067 to 5.080]
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.049, 95% CI 2-sided [1.317 to 3.210]
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.097, 95% CI 2-sided [1.994 to 4.858]
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.984, 95% CI 2-sided [1.280 to 3.097]
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.062, 95% CI 2-sided [1.977 to 4.788]
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.748, 95% CI 2-sided [1.774 to 4.294]
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.379, 95% CI 2-sided [1.536 to 3.712]
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.051, 95% CI 2-sided [1.329 to 3.186]
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.701, 95% CI 2-sided [1.750 to 4.204]
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.725, 95% CI 2-sided [1.742 to 4.306]
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.921, 95% CI 2-sided [2.505 to 6.214]
Statistical Analysis 21: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.104, 95% CI 2-sided [1.363 to 3.270]
Statistical Analysis 22: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.953, 95% CI 2-sided [1.912 to 4.602]
Statistical Analysis 23: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 12; Test type: Superiority; p = 0.005, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.894, 95% CI 2-sided [1.220 to 2.961]
Statistical Analysis 24: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.156, 95% CI 2-sided [2.035 to 4.944]

10. Secondary Outcome: Number of Participants With Mean Percent Reduction of 100% in The Mean Frequency of Moderate, and Severe VMS From Baseline to Each Study Week Up to Week 12
Description: The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. A daily frequency per week was derived by taking the mean of the data over 7 days. Moderate VMS was defined as sensation of heat with sweating/dampness, but participant was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). Baseline was the average number of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization. Participant has 100% reduction from baseline to each post baseline week for the frequency of moderate to severe VMS.
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: FAS Population
Measure: Number; unit: Participants
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 175 | 173 | 174
Participants
  Week 1 | 0 | 0 | 0
  Week 2 | 1 | 3 | 4
  Week 3 | 1 | 6 | 5
  Week 4 | 5 | 6 | 8
  Week 5 | 2 | 10 | 6
  Week 6 | 2 | 8 | 10
  Week 7 | 2 | 13 | 13
  Week 8 | 2 | 10 | 14
  Week 9 | 5 | 15 | 16
  Week 10 | 7 | 17 | 18
  Week 11 | 10 | 16 | 19
  Week 12 | 6 | 12 | 18
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p = 0.322, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.158, 95% CI 2-sided [0.398 to 64.304]
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p = 0.225, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.925, 95% CI 2-sided [0.569 to 77.353]
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p = 0.089, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 6.334, 95% CI 2-sided [1.064 to 120.422]
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p = 0.143, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 5.026, 95% CI 2-sided [0.797 to 96.916]
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 4; Test type: Superiority; p = 0.711, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.257, 95% CI 2-sided [0.370 to 4.468]
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 4; Test type: Superiority; p = 0.441, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.570, 95% CI 2-sided [0.508 to 5.328]
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p = 0.032, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 5.351, 95% CI 2-sided [1.383 to 35.172]
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p = 0.175, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.059, 95% CI 2-sided [0.693 to 21.086]
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p = 0.071, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 4.225, 95% CI 2-sided [1.039 to 28.290]
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p = 0.035, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 5.220, 95% CI 2-sided [1.348 to 34.323]
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p = 0.011, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 7.064, 95% CI 2-sided [1.912 to 45.640]
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p = 0.012, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 6.949, 95% CI 2-sided [1.881 to 44.892]
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p = 0.032, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 5.344, 95% CI 2-sided [1.381 to 35.134]
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p = 0.008, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 7.514, 95% CI 2-sided [2.055 to 48.354]
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p = 0.026, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.238, 95% CI 2-sided [1.222 to 10.148]
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p = 0.019, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.438, 95% CI 2-sided [1.311 to 10.714]
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p = 0.037, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.626, 95% CI 2-sided [1.101 to 6.951]
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p = 0.027, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.758, 95% CI 2-sided [1.167 to 7.263]
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p = 0.210, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.690, 95% CI 2-sided [0.753 to 3.968]
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p = 0.087, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.010, 95% CI 2-sided [0.923 to 4.634]
Statistical Analysis 21: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 12; Test type: Superiority; p = 0.148, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.100, 95% CI 2-sided [0.795 to 6.157]
Statistical Analysis 22: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 12; Test type: Superiority; p = 0.015, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.262, 95% CI 2-sided [1.329 to 9.194]

11. Secondary Outcome: Number of Participants in Each Category of Patient's Global Impression of Change (PGIC) in VMS at Each Visit
Description: The PGI is comprised of 2 companion 1-item PRO measures analogous to the Clinical Global Impression (CGI) scales. These measures provide brief, stand-alone global assessments prior to and after initiating a study medication. Patient-perceived change from the initiation of treatment (PGI-C)-VMS is used to evaluate meaningful within-person changes over time in VMS. This measure provides patient-perceived change from the initiation of treatment.
  The PGI-C VMS asks: "Compared to the beginning of this study, how would you rate your HFs/night sweats now?" Subject ratings range from (1) much better to (7) much worse. Participant ratings range from 1=much better, 2= moderately better, 3= a little better, 4= no change, 5= a little worse, 6= moderately worse, 7= much worse.
Time Frame: Weeks 4, 12, 16, 20, 24, 28, 32, 36, 40, 48, 52 of fezolinetant exposure (weeks 16, 24, 28, 32, 36, 40, 44, 48 and 52 for arms Placebo/Fezolinetant 30 mg and Placebo/Fezolinetant 45 mg)
Population: FAS population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Number analyzed (Participants) | 160 | 150 | 160 | 68 | 70
Participants
  Week 4: Much better: number analyzed (Participants) | 160 | 150 | 160 | 0 | 1
  Week 4: Much better | 32 | 50 | 72 |  | 1
  Week 4: Moderately better: number analyzed (Participants) | 160 | 150 | 160 | 0 | 1
  Week 4: Moderately better | 21 | 33 | 24 |  | 0
  Week 4: A little better: number analyzed (Participants) | 160 | 150 | 160 | 0 | 1
  Week 4: A little better | 44 | 42 | 35 |  | 0
  Week 4: No change: number analyzed (Participants) | 160 | 150 | 160 | 0 | 1
  Week 4: No change | 55 | 23 | 28 |  | 0
  Week 4: A little worse: number analyzed (Participants) | 160 | 150 | 160 | 0 | 1
  Week 4: A little worse | 1 | 1 | 0 |  | 0
  Week 4: Moderately worse: number analyzed (Participants) | 160 | 150 | 160 | 0 | 1
  Week 4: Moderately worse | 1 | 1 | 1 |  | 0
  Week 4: Much worse: number analyzed (Participants) | 160 | 150 | 160 | 0 | 1
  Week 4: Much worse | 6 | 0 | 0 |  | 0
  Week 12: Much better: number analyzed (Participants) | 149 | 136 | 157 | 68 | 70
  Week 12: Much better | 35 | 50 | 74 | 31 | 44
  Week 12: Moderately better: number analyzed (Participants) | 149 | 136 | 157 | 68 | 70
  Week 12: Moderately better | 24 | 24 | 30 | 14 | 16
  Week 12: A little better: number analyzed (Participants) | 149 | 136 | 157 | 68 | 70
  Week 12: A little better | 40 | 41 | 35 | 16 | 8
  Week 12: No change: number analyzed (Participants) | 149 | 136 | 157 | 68 | 70
  Week 12: No change | 37 | 19 | 11 | 4 | 2
  Week 12: A little worse: number analyzed (Participants) | 149 | 136 | 157 | 68 | 70
  Week 12: A little worse | 6 | 1 | 2 | 1 | 0
  Week 12: Moderately worse: number analyzed (Participants) | 149 | 136 | 157 | 68 | 70
  Week 12: Moderately worse | 4 | 1 | 4 | 2 | 0
  Week 12: Much worse: number analyzed (Participants) | 149 | 136 | 157 | 68 | 70
  Week 12: Much worse | 3 | 0 | 1 | 0 | 0
  Week 16: Much better: number analyzed (Participants) | 0 | 5 | 4 | 1 | 0
  Week 16: Much better |  | 1 | 2 | 0 |
  Week 16: Moderately better: number analyzed (Participants) | 0 | 5 | 4 | 1 | 0
  Week 16: Moderately better |  | 2 | 1 | 0 |
  Week 16: A little better: number analyzed (Participants) | 0 | 5 | 4 | 1 | 0
  Week 16: A little better |  | 1 | 1 | 1 |
  Week 16: No change: number analyzed (Participants) | 0 | 5 | 4 | 1 | 0
  Week 16: No change |  | 1 | 0 | 0 |
  Week 16: A little worse: number analyzed (Participants) | 0 | 5 | 4 | 1 | 0
  Week 16: A little worse |  | 0 | 0 | 0 |
  Week 16: Moderately worse: number analyzed (Participants) | 0 | 5 | 4 | 1 | 0
  Week 16: Moderately worse |  | 0 | 0 | 0 |
  Week 16: Much worse: number analyzed (Participants) | 0 | 5 | 4 | 1 | 0
  Week 16: Much worse |  | 0 | 0 | 0 |
  Week 20: Much better: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  Week 20: Much better |  | 1 | 1 |  |
  Week 20: Moderately better: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  Week 20: Moderately better |  | 1 | 0 |  |
  Week 20: A little better: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  Week 20: A little better |  | 0 | 2 |  |
  Week 20: No change: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  Week 20: No change |  | 1 | 1 |  |
  Week 20: A little worse: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  Week 20: A little worse |  | 0 | 0 |  |
  Week 20: Moderately worse: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  Week 20: Moderately worse |  | 0 | 0 |  |
  Week 20: Much worse: number analyzed (Participants) | 0 | 3 | 4 | 0 | 0
  Week 20: Much worse |  | 0 | 0 |  |
  Week 24: Much better: number analyzed (Participants) | 0 | 127 | 148 | 0 | 0
  Week 24: Much better |  | 55 | 81 |  |
  Week 24: Moderately better: number analyzed (Participants) | 0 | 127 | 148 | 0 | 0
  Week 24: Moderately better |  | 27 | 30 |  |
  Week 24: A little better: number analyzed (Participants) | 0 | 127 | 148 | 0 | 0
  Week 24: A little better |  | 34 | 27 |  |
  Week 24: No change: number analyzed (Participants) | 0 | 127 | 148 | 0 | 0
  Week 24: No change |  | 10 | 6 |  |
  Week 24: A little worse: number analyzed (Participants) | 0 | 127 | 148 | 0 | 0
  Week 24: A little worse |  | 0 | 1 |  |
  Week 24: Moderately worse: number analyzed (Participants) | 0 | 127 | 148 | 0 | 0
  Week 24: Moderately worse |  | 1 | 2 |  |
  Week 24: Much worse: number analyzed (Participants) | 0 | 127 | 148 | 0 | 0
  Week 24: Much worse |  | 0 | 1 |  |
  Week 28: Much better: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Week 28: Much better |  | 0 | 1 |  |
  Week 28: Moderately better: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Week 28: Moderately better |  | 0 | 0 |  |
  Week 28: A little better: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Week 28: A little better |  | 0 | 0 |  |
  Week 28: No change: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Week 28: No change |  | 0 | 0 |  |
  Week 28: A little worse: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Week 28: A little worse |  | 0 | 0 |  |
  Week 28: Moderately worse: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Week 28: Moderately worse |  | 0 | 0 |  |
  Week 28: Much worse: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Week 28: Much worse |  | 0 | 0 |  |
  Week 32: Much better: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: Much better |  |  | 0 |  |
  Week 32: Moderately better: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: Moderately better |  |  | 1 |  |
  Week 32: A little better: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: A little better |  |  | 0 |  |
  Week 32: No change: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: No change |  |  | 0 |  |
  Week 32: A little worse: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: A little worse |  |  | 0 |  |
  Week 32: Moderately worse: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: Moderately worse |  |  | 0 |  |
  Week 32: Much worse: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: Much worse |  |  | 0 |  |
  Week 36: Much better: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Week 36: Much better |  |  | 0 | 0 |
  Week 36: Moderately better: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Week 36: Moderately better |  |  | 1 | 1 |
  Week 36: A little better: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Week 36: A little better |  |  | 0 | 0 |
  Week 36: No change: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Week 36: No change |  |  | 0 | 0 |
  Week 36: A little worse: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Week 36: A little worse |  |  | 0 | 0 |
  Week 36: Moderately worse: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Week 36: Moderately worse |  |  | 0 | 0 |
  Week 36: Much worse: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Week 36: Much worse |  |  | 0 | 0 |
  Week 40: Much better: number analyzed (Participants) | 0 | 2 | 0 | 55 | 63
  Week 40: Much better |  | 0 |  | 33 | 39
  Week 40: Moderately better: number analyzed (Participants) | 0 | 2 | 0 | 55 | 63
  Week 40: Moderately better |  | 2 |  | 8 | 12
  Week 40: A little better: number analyzed (Participants) | 0 | 2 | 0 | 55 | 63
  Week 40: A little better |  | 0 |  | 6 | 10
  Week 40: No change: number analyzed (Participants) | 0 | 2 | 0 | 55 | 63
  Week 40: No change |  | 0 |  | 6 | 1
  Week 40: A little worse: number analyzed (Participants) | 0 | 2 | 0 | 55 | 63
  Week 40: A little worse |  | 0 |  | 2 | 1
  Week 40: Moderately worse: number analyzed (Participants) | 0 | 2 | 0 | 55 | 63
  Week 40: Moderately worse |  | 0 |  | 0 | 0
  Week 40: Much worse: number analyzed (Participants) | 0 | 2 | 0 | 55 | 63
  Week 40: Much worse |  | 0 |  | 0 | 0
  Week 48: Much better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 48: Much better |  | 0 |  |  |
  Week 48: Moderately better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 48: Moderately better |  | 1 |  |  |
  Week 48: A little better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 48: A little better |  | 1 |  |  |
  Week 48: No change: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 48: No change |  | 0 |  |  |
  Week 48: A little worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 48: A little worse |  | 0 |  |  |
  Week 48: Moderately worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 48: Moderately worse |  | 0 |  |  |
  Week 48: Much worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 48: Much worse |  | 0 |  |  |
  Week 52: Much better: number analyzed (Participants) | 0 | 111 | 127 | 0 | 0
  Week 52: Much better |  | 56 | 71 |  |
  Week 52: Moderately better: number analyzed (Participants) | 0 | 111 | 127 | 0 | 0
  Week 52: Moderately better |  | 26 | 30 |  |
  Week 52: A little better: number analyzed (Participants) | 0 | 111 | 127 | 0 | 0
  Week 52: A little better |  | 23 | 15 |  |
  Week 52: No change: number analyzed (Participants) | 0 | 111 | 127 | 0 | 0
  Week 52: No change |  | 6 | 8 |  |
  Week 52: A little worse: number analyzed (Participants) | 0 | 111 | 127 | 0 | 0
  Week 52: A little worse |  | 0 | 1 |  |
  Week 52: Moderately worse: number analyzed (Participants) | 0 | 111 | 127 | 0 | 0
  Week 52: Moderately worse |  | 0 | 1 |  |
  Week 52: Much worse: number analyzed (Participants) | 0 | 111 | 127 | 0 | 0
  Week 52: Much worse |  | 0 | 1 |  |

12. Secondary Outcome: Change From Baseline in The Mean Frequency of Moderate, and Severe VMS at Week 24
Description: as for outcome 1
Time Frame: Baseline and 24 weeks of fezolinetant exposure (week 36 for arms Placebo/Fezolinetanat 30 mg and Placebo/Fezolinetant 45 mg)
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: VMS per day
Arm/Group | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Number analyzed (Participants) | 121 | 138 | 60 | 62
VMS per day | -7.15 (6.02) | -7.32 (4.58) | -6.89 (3.67) | -7.32 (4.53)

13. Secondary Outcome: Change From Baseline in The Mean Severity of Moderate, and Severe VMS at Week 24
Description: as for outcome 3
Time Frame: as for outcome 12
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Number analyzed (Participants) | 121 | 138 | 60 | 62
Score on a scale | -0.75 (0.82) | -0.77 (0.90) | -0.78 (0.80) | -0.76 (0.89)

14. Secondary Outcome: Number of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a participant administered a study drug, & which does not necessarily have to have a causal relationship with treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with use of a medicinal product (mp) whether or not considered related to the mp. An AE is considered "serious" if it results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires inpatient hospitalization or leads to prolongation of hospitalization, hospitalization for treatment/observation/examination caused by AE is to be considered as serious, discontinuation due to increases in liver enzymes, other medically important events. TEAE was defined as an AE observed from first dose date up to 21 days after last dose.
Time Frame: From first dose date up to 21 days after last dose (to 55 weeks)
Population: Safety population included all randomized participants who took at least 1 dose of study intervention. A participant erroneously receiving a treatment different from their randomized treatment was assigned to the treatment group that the participant received as first dose.
Measure: Number; unit: Participants
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Number analyzed (Participants) | 175 | 174 | 173 | 76 | 76
Participants
  TEAE | 78 | 108 | 115 | 48 | 37
  Drug-Related TEAE | 22 | 20 | 21 | 6 | 2
  Serious TEAE | 1 | 7 | 8 | 3 | 2
  Drug-Related Serious TEAE | 0 | 2 | 0 | 0 | 0
  TEAE Leading to Death | 0 | 0 | 0 | 0 | 0
  Drug-Related TEAE Leading to Death | 0 | 0 | 0 | 0 | 0
  TEAE Leading to Withdrawal of Treatment | 9 | 13 | 8 | 2 | 1
  Drug-Related TEAE Leading to Withdrawal of Treatment | 7 | 7 | 5 | 0 | 1
  Death | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose date up to 21 days after last dose (up to 55 weeks)
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/174 | 0/173 | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/175 | 7/174 | 8/173 | 3/76 | 2/76
Other Adverse Events (participants affected / at risk) | 24/175 | 38/174 | 45/173 | 18/76 | 14/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Period: Placebo (N=175) | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg (N=174) | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg (N=173) | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg (N=76) | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg (N=76)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apocrine breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Period: Placebo (N=175) | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg (N=174) | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg (N=173) | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg (N=76) | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg (N=76)
COVID-19 (Infections and infestations) | 0 (0) | 9 (9) | 11 (11) | 4 (4) | 6 (6)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (6) | 9 (9) | 2 (2) | 1 (2)
Alanine aminotransferase increased (Investigations) | 4 (4) | 8 (9) | 10 (13) | 2 (2) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 6 (6) | 6 (6) | 5 (8) | 5 (11) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 10 (15) | 8 (14) | 2 (4) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 6 (8) | 7 (12) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 13 (14) | 11 (17) | 14 (15) | 3 (5) | 5 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT04003155/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04003155/SAP_001.pdf